CLINICAL TRIAL: NCT03261869
Title: EFFICACY OF ICE PACK THERAPY AFTER IMPACTED THIRD MOLAR SURGERY: A RANDOMIZED CONTROLLED CLINICAL TRIAL
Brief Title: EFFICACY OF ICE PACK THERAPY AFTER IMPACTED THIRD MOLAR SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nurettin Diker, Research Assistant at deparment of oral and maxillofacial surgery, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: D-KA 15/07
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: Ice pack therapy, third molar surgery, swelling, pain, trismus
MeSH Terms: conditions — Pain; Trismus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold application (Experimental): Cold applied after extraction of third molar tooth.
  Interventions: Other: Cold application
- No Cold application (No Intervention): Cold application is not advised after extraction of third molar tooth

INTERVENTIONS:
Other: Cold application
  Arms: Cold application

SUMMARY:
this study evaluates the effect of cold application after impacted third molar extractions. Patients have bilateral impacted third molar tooth included in this study. Patients do not applied cold after extraction of third molar on one side and applied cold cold after extraction of third molar on the other side.

DETAILED DESCRIPTION:
Extraction of impacted teeth causes a trauma which results in an inflammatory response. Some postoperative symptoms may occur such as edema, pain, limitations in mouth opening and dysfunction as a consequence of the wisdom tooth extraction surgery.

Local cold application reduces the magnitude of postoperative symptoms. The physiological effects of cold application are as follows: vasoconstriction of blood vessels, blood flow to the region decreases, edema and inflammation decreases, slowdown in cell metabolism and a decrease in local oxygen demand due to the vasoconstriction effect of the cold. Cold therapy also induces muscle constriction which reduces muscle stress, pain and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral bony mandibular third molar impactions
* Has no systemic disease

Exclusion Criteria:

* Different Pell-Gregory classification of impacted teeth
* Previous or current gastric ulcer
* Allergies or hypersensitivities to any common medications
* pregnant or breastfeeding patients

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Post operative Visual Analogue Scale Scores | pre-operative-postoperative 7th day
Post operative facial swelling | pre-operative-postoperative 7th day
Post-operative mouth opening | pre-operative-postoperative 7th day

SECONDARY OUTCOMES:
Complications after impacted third molar removal | pre-operative-postoperative 7th day

IPD SHARING:
Plan to Share IPD: No